CLINICAL TRIAL: NCT00189098
Title: Effectiveness of Sulfamethoxazole-trimethoprim in the Treatment of Chronic Otitis Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Health Care Insurance Board (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VAZ 01-235
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Otitis Media
MeSH Terms: interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Sulfamethoxazole-trimethoprim (Active Comparator)
  Interventions: Drug: Sulfamethoxazole-trimethoprim

INTERVENTIONS:
Drug: Sulfamethoxazole-trimethoprim — 18 mg/kg, two times a day
  Arms: Sulfamethoxazole-trimethoprim
Drug: Placebo
  Arms: placebo

SUMMARY:
Chronic suppurative otitis media is one of the most common chronic infections in children worldwide. Symptoms include otorrhea, otalgia and hearing loss. In many countries, it is treated primarily with antibiotics; in other countries such as the Netherlands a surgical approach, such as a tonsillectomy, adenoidectomy, placement or removal of tympanostomy tubes or a tympanomastoidectomy is preferred. There is however, no agreement on the management of this disease.

The purpose of this study is to determine the effectiveness of treatment with sulfamethoxazole-trimethoprim for 6-12 weeks in children suffering from chronic otitis media and otorrhea.

DETAILED DESCRIPTION:
Chronic suppurative otitis media is one of the most common chronic infections in children worldwide. Symptoms include otorrhea, otalgia and hearing loss. In many countries it is treated primarily with antibiotics; in other countries such as the Netherlands a surgical approach, such as a tonsillectomy, adenoidectomy, placement or removal of tympanostomy tubes or a tympanomastoidectomy is preferred. There is however, no agreement on the management of this disease.

Co-trimoxazole is an inexpensive antibiotic and tolerated well by children, also when long treatment regimens or prophylaxis is necessary. A previously performed retrospective study of 48 children who were referred to the pediatric department of otorhinolaryngology in the UMC Utrecht because of "therapeutic resistant" otorrhea showed promising results; after 3 months follow-up, 52% of the patients were otorrhea free, 25% had otorrhea incidentally and 23% showed no signs of improvement. Therefore, the treatment of chronic otitis media with sulfamethoxazole-trimethoprim for a minimum of six weeks is promising and might be a good alternative to surgical treatment.

The purpose of this study is to determine the effectiveness of treatment with sulfamethoxazole-trimethoprim during 6-12 weeks in children with chronic otitis media and otorrhea for more than 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age between 1 and 12 years
* otorrhea for more than 3 months

Exclusion Criteria:

* cholesteatoma
* known immune deficiency other than IgA or IgG2
* Down's syndrome
* craniofacial anomalies
* cystic fibrosis
* immotile cilia syndrome
* allergy to sulfamethoxazole-trimethoprim
* continuous use of sulfamethoxazole-trimethoprim for more than six weeks in the past six months

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2003-02; Primary Completion 2006-06 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne GM Schilder, MD, PhD, Study Director — University Medical Centre Utrecht, Department of Pediatric Otorhinolaryngology
Locations (1):
- Wilhelmina Children Hospital, University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] van der Veen EL, Rovers MM, Albers FW, Sanders EA, Schilder AG. Effectiveness of trimethoprim/sulfamethoxazole for children with chronic active otitis media: a randomized, placebo-controlled trial. Pediatrics. 2007 May;119(5):897-904. doi: 10.1542/peds.2006-2787. PMID 17473089
- [Derived] van der Veen EL, Schilder AG, Timmers TK, Rovers MM, Fluit AC, Bonten MJ, Leverstein-van Hall MA. Effect of long-term trimethoprim/sulfamethoxazole treatment on resistance and integron prevalence in the intestinal flora: a randomized, double-blind, placebo-controlled trial in children. J Antimicrob Chemother. 2009 May;63(5):1011-6. doi: 10.1093/jac/dkp050. Epub 2009 Mar 18. PMID 19297377

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between February 2003 and June 2006. Otorhinolaryngologists and paediatricians from all over the Netherlands referred potential participants, i.e. children with COM that had failed conventional management with topical medications and/or short term systemic antibiotics
Groups:
- Placebo: Children assigned to the placebo group received two times a day a placebo for 6 to 12 weeks. The placebo was a blinded suspension with an identical taste, bottle and fluid appearance as the sulfamethoxazole-trimethoprim suspension. When at the first control visit after 6 weeks otorrhea was found to be present in either ear, the study medication was continued for another 6 weeks. The study medication was discontinued if both ears were found to be free from otorrhea and parents confirmed that they had seen no signs of otorrhea during the previous week. Parents were instructed to start the study medication again if symptoms of otorrhea recurred between the follow-up visits at 6 and 12 weeks. At inclusion and if otorrhea was present at 6 and 12 weeks follow-up, antibiotic with corticosteroid eardrops were prescribed in addition to the study medication for 7 to 10 days. After 12 weeks follow-up the study medication was discontinued irrespective of the presence or absence of otorrhea.
- Sulfamethoxazole-trimethoprim: Children assigned to the Sulfamethoxazole-trimethoprim group received Sulfamethoxazole-trimethoprim orally (18mg/kg two times a day) for 6 to 12 weeks. When at the first control visit after 6 weeks otorrhea was found to be present in either ear, the study medication was continued for another 6 weeks. The study medication was discontinued if both ears were found to be free from otorrhea and parents confirmed that they had seen no signs of otorrhea during the previous week. Parents were instructed to start the study medication again if symptoms of otorrhea recurred between the follow-up visits at 6 and 12 weeks. At inclusion and if otorrhea was present at 6 and 12 weeks follow-up, antibiotic with corticosteroid eardrops were prescribed in addition to the study medication for 7 to 10 days. After 12 weeks follow-up the study medication was discontinued irrespective of the presence or absence of otorrhea.
Period: Overall Study
Arm/Group | Placebo | Sulfamethoxazole-trimethoprim
Started | 51 | 50
Completed | 46 | 44
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sulfamethoxazole-trimethoprim | Total
Number analyzed (Participants) | 51 | 50 | 101
Age Continuous [Median (Full Range); unit: months] | 51 [15 to 143] | 48 [12 to 144] | 50 [12 to 144]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Otomicroscopic Signs of Otorrhea in Either Ear
Description: The primary endpoint was otomicroscopic signs of otorrhea in either ear in the presence of a tympanostomy tube or tympanic membrane perforation at 6 and 12 weeks and 1 year follow-up. At these follow-up moments the participants were checked for the presence of otorrhea using an otomicroscope.
Time Frame: 6, 12 weeks and 1 year follow-up.
Population: intention to treat
Measure: Number; unit: participants
Groups:
- Sulfamethoxazole-trimethoprim: The children in this group received Sulfamethoxazole-trimethoprim orally (18 mg/kg, two times a day) for 6 to 12 weeks.
- Placebo: The children in this group received placebo orally two times a day for 6 to 12 weeks.
Arm/Group | Sulfamethoxazole-trimethoprim | Placebo
Number analyzed (Participants) | 44 | 46
participants
  At 6 weeks | 13 | 27
  At 12 weeks | 15 | 23
  At 12 months | 11 | 9
Statistical Analysis 1: Comparison: Sulfamethoxazole-trimethoprim vs Placebo; Assuming a spontaneous recovery of 25% and a treatment effect of TMP-SMX of 50% (based on a retrospective study of children treated with TMP-SMX for COM at our hospital), and taking α=0.05 and a power of 0.80, we calculated that each group should consist of 50 children. Rate differences with 95% confidence intervals were calculated at the three control visits to compare both groups for the outcome measures; Test type: Superiority or Other; risk differences (RD); Risk Difference (RD) = -25, 95% CI 2-sided [-44 to -6] — Risk difference and 95% confidence intervals reported for 6 weeks follow-up
Statistical Analysis 2: Comparison: Sulfamethoxazole-trimethoprim vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; risk difference (RD); Risk Difference (RD) = -15, 95% CI 2-sided [-34 to 4] — Risk difference and confidence interval reported for 12 week follow-up
Statistical Analysis 3: Comparison: Sulfamethoxazole-trimethoprim vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; risk difference (RD); Risk Difference (RD) = 5, 95% CI 2-sided [-12 to 22] — Risk difference and confidence interval reported for 1 year follow-up

2. Secondary Outcome: Number of Patients Who Used Additional Antibiotic Eardrops Between 6 to 12 Week Follow-up
Description: Parents kept a diary of study medication and additional medication used for their child's' ear disease, including eardrops. These data were collected at the follow-up visits.
Time Frame: Between 6 to12 week follow up
Population: Parents kept a diary of study medication and additional medication used for their child's' ear disease, including eardrops. These data were collected at the follow-up visits. Some parents did not fill in the required forms and these were excluded in this analysis. Therefore number of participants analyzed differ from the flow-chart.
Measure: Number; unit: participants
Arm/Group | Sulfamethoxazole-trimethoprim | Placebo
Number analyzed (Participants) | 38 | 39
participants | 21 | 26
Statistical Analysis 1: Comparison: Sulfamethoxazole-trimethoprim vs Placebo; Test type: Superiority or Other; rate differences (95%CI intervals); Risk Difference (RD) = -12, 95% CI 2-sided [-34 to 10] — Risk difference and confidence interval reported for eardrop usage between 6 and 12 weeks follow-up

3. Secondary Outcome: Number of Patients Who Used Additional Antibiotic Eardrops Between 12 Weeks to 1 Year Follow-up
Description: as for outcome 2
Time Frame: between 12 weeks to 1 year follow-up
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Sulfamethoxazole-trimethoprim | Placebo
Number analyzed (Participants) | 37 | 38
participants | 29 | 31
Statistical Analysis 1: Comparison: Sulfamethoxazole-trimethoprim vs Placebo; Test type: Superiority or Other; rate difference (RD); Risk Difference (RD) = -4, 95% CI 2-sided [-22 to 14] — Risk difference and confidence interval reported for eardrop usage between 12 weeks and 1 year follow-up

4. Secondary Outcome: Number of Patients Who Used Systemic Antibiotics Other Than the Study Medication Between 6 and 12 Weeks Follow-up.
Description: Parents kept a diary of study medication and additional medication used for their child's' ear disease, including additional use of systemic antibiotics other than the study medication. These data were collected at the follow-up visits.
Time Frame: between 6 and 12 weeks follow-up
Population: Parents kept a diary of study medication and additional medication used for their child's' ear disease, including additional use of systemic antibiotics other than the study medication. These data were collected at the follow-up visits. Some parents did not fill in the required forms and these were excluded in this analysis.
Measure: Number; unit: participants
Arm/Group | Sulfamethoxazole-trimethoprim | Placebo
Number analyzed (Participants) | 38 | 39
participants | 4 | 7
Statistical Analysis 1: Comparison: Sulfamethoxazole-trimethoprim vs Placebo; Test type: Superiority or Other; Rate differences (95%CI interval); Risk Difference (RD) = -7, 95% CI 2-sided [-23 to 9] — Risk difference and confidence interval reported for the use of additional systemic antibiotics other than the study medication between 6 to 12 weeks follow-up

5. Secondary Outcome: Number of Patients Who Used Systemic Antibiotics Other Than the Study Medication Between 12 Weeks and 1 Year Follow-up.
Description: as for outcome 4
Time Frame: between 12 weeks and 1 year follow-up
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Sulfamethoxazole-trimethoprim | Placebo
Number analyzed (Participants) | 37 | 38
participants | 23 | 18
Statistical Analysis 1: Comparison: Sulfamethoxazole-trimethoprim vs Placebo; Test type: Superiority or Other; Rate difference (RD); Risk Difference (RD) = 15, 95% CI 2-sided [-7 to 37] — Risk difference and confidence interval reported for the use of additional systemic antibiotics other than the study medication between 12 weeks and 1 year follow-up

6. Secondary Outcome: Number of Patients Who Underwent Ear Nose and Throat Surgery Between 12 Weeks and 1 Year Follow-up.
Description: After 12 weeks follow-up irrespective of the presence or absence of otorrhea the study medication was discontinued. After the first 12 weeks local otorhinolaryngologists and paediatricians were free to manage symptoms of otorrhea according to their regular practice. Parents kept a diary between 12 weeks and 1 year follow-up where Ear Nose and Throat Surgery was noted. This outcome describes the number of patients who underwent Ear Nose and Throat Surgery between 12 weeks and 1 year follow-up.
Time Frame: between 12 weeks and 1 year follow-up
Measure: Number; unit: participants
Arm/Group | Sulfamethoxazole-trimethoprim | Placebo
Number analyzed (Participants) | 44 | 46
participants | 13 | 11
Statistical Analysis 1: Comparison: Sulfamethoxazole-trimethoprim vs Placebo; Test type: Superiority or Other; Rate differences (95%CI intervals); Risk Difference (RD) = 6, 95% CI 2-sided [-12 to 24] — Risk difference and confidence interval reported for participants who underwent Ear Nose and Throat Surgery between 12 weeks and 1 year follow-up

ADVERSE EVENTS:
Time Frame: During the first 12 weeks
Description: Using diaries
Arm/Group | Sulfamethoxazole-trimethoprim | Placebo
Serious Adverse Events (participants affected / at risk) | 1/50 | 1/51
Other Adverse Events (participants affected / at risk) | 4/50 | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulfamethoxazole-trimethoprim (N=50) | Placebo (N=51)
Mastoiditis (Ear and labyrinth disorders) | 1 (1) | 1 (1) — Mastoiditis was measured by using the diaries and hospital admissions
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulfamethoxazole-trimethoprim (N=50) | Placebo (N=51)
vomiting or diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
skinrash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No